CLINICAL TRIAL: NCT03267862
Title: Scleral Response to Intraocular Pressure (IOP)
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: NA_00090957
Record Dates: First submitted 2017-08-29; First posted 2017-08-30 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Glaucoma, Open-Angle
Keywords: biomarker
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: there was no intervention — patients were observed during routine care on separate times when their eye pressure was different on one day from another.

SUMMARY:
The study evaluated changes in the depth of the lamina cribrosa at different eye pressures.

DETAILED DESCRIPTION:
Participants were glaucoma patients who during routine care were observed at different eye pressures. Images taken with an optical device that is routinely used in such patients were analysed.

ELIGIBILITY:
Inclusion Criteria:

* glaucoma patients

Exclusion Criteria:

* non-glaucoma patients

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: glaucoma patients presenting for routine care
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2014-09-17 (Actual); Primary Completion 2017-08-29 (Actual); Study Completion 2017-08-29 (Actual)

PRIMARY OUTCOMES:
Anterior lamina cribrosa depth change | Up to 2 months
  Position of anterior lamina observed by optical coherence tomography (OCT) imaging. Measured in micrometers (um).

IPD SHARING:
Plan to Share IPD: Undecided
deidentified study data could be shared at this time